CLINICAL TRIAL: NCT01965665
Title: Advancing the Standard of Care for Pin Site Care: Prospective Single Center Study Using Medihoney HCS
Brief Title: Advancing the Standard of Care for Pin Site Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00046972
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus; Open Reduction External Fixation
Keywords: Diabetes; Surgical Intervention; Honey
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Medihoney HCS dressing (Experimental): weekly Medihoney pin site care until frame removal. Standard size dressings and application technique will be used at each pin site with prefabricated materials.
  Interventions: Device: MediHoney HCS dressing

INTERVENTIONS:
Device: MediHoney HCS dressing

SUMMARY:
The purpose of this study is to prospectively evaluate the effect of Active Leptospermum honey utilizing the MediHoney HCS dressing, on the occurrence of PIN site infections, and also to see if the use of MediHoney HCS reduces the frequency of dressing changes compared to published reports of routine standard pin site care.

DETAILED DESCRIPTION:
Up to 20 Diabetic Mellitus patients undergoing Open Reduction External Fixation (OREF) for foot and/or ankle fusions, fracture repair, or osteotomy will be enrolled to receive weekly Medihoney pin site care until frame removal. Standard size dressings and application technique will be used at each pin site with prefabricated materials. No procedures, tests or interventions will be performed exclusively for research purposes or more frequently than the standard of care. Upon completion of the study, pin sites sepsis rates will be compared to published reports for standard pin site care.

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent has been obtained from the subject.
* Subject is able and willing to comply with study procedures.
* Subject is 18 years of age or older.
* Type I or II Diabetes
* Albumin >2.5
* A1C<12 or average fasting levels <200
* ABI > .6 or biphasic pedal vessels by Doppler
* Charcot arthropathy of lower extremity

  * Foot/ankle deformity
  * Foot/ankle fracture
* Subject will undergo an Open Reduction with External Fixation (OREF).

Exclusion Criteria:

* A1C > 12
* ABI < .6 or monophasic pedal pulses on Doppler
* Recent (<2 months) or ongoing bone infection based on radiograph or scan
* Cellulitis of lower extremity within the last 2 months based on clinical exam and/or laboratory markers
* Honey or honey based allergy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kerzner, DPM, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center/Duke South Clinics/3J, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Medihoney HCS Dressing: weekly Medihoney pin site care until frame removal. Standard size dressings and application technique will be used at each pin site with prefabricated materials.
  MediHoney HCS dressing
Period: Overall Study
Arm/Group | Medihoney HCS Dressing
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Medihoney HCS Dressing
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Pin Sites
Description: total number of pin sites for all patients enrolled
Time Frame: Day of surgical intervention approximately 3hrs.
Measure: Number; unit: total number of pin sites
Arm/Group | Medihoney HCS Dressing
Number analyzed (Participants) | 19
total number of pin sites | 244

2. Primary Outcome: Number of Patients With Pin Site Infection
Description: Patients will be assessed weekly for pin site infection up until frame removal.
Time Frame: weekly from baseline until frame removal, up to 16 weeks
Measure: Number; unit: participants
Arm/Group | Medihoney HCS Dressing
Number analyzed (Participants) | 19
participants | 3

3. Primary Outcome: Change in Sepsis Rate
Description: Patients will be assessed weekly for sepsis or until frame is removed.
Time Frame: weekly from baseline until frame removal, up to 16 weeks
Population: Data not collected
Arm/Group | Medihoney HCS Dressing
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: baseline until frame removal, up to 16 weeks
Arm/Group | Medihoney HCS Dressing
Serious Adverse Events (participants affected / at risk) | 1/19
Other Adverse Events (participants affected / at risk) | 1/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medihoney HCS Dressing (N=19)
GI infection (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medihoney HCS Dressing (N=19)
osteotomy site infection (not pin site) (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes